CLINICAL TRIAL: NCT06633588
Title: Surgical Prophylaxis: Assessing Decolonization Efficacy of Polyhexanide Versus Mupirocin and Chlorhexidine in Decolonizing Staphylococcus Aureus Preoperatively in Elective Spine Surgery (SPADE): A Pilot Randomized Controlled Trial
Brief Title: Decolonization Efficacy of Polyhexanide vs. Mupirocin
Acronym: SPADE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-08
Record Dates: First submitted 2024-09-19; First posted 2024-10-09 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Staphylococcus Aureus; Colonization, Asymptomatic
Keywords: Staphylococcus aureus colonization; Spinal surgery; decolonization
MeSH Terms: conditions — Staphylococcal Infections; Asymptomatic Infections | interventions — polihexanide; Mupirocin; Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyhexanide (Experimental)
  Interventions: Drug: Polyhexanide
- Mupirocin and Chlorhexidine (Active Comparator)
  Interventions: Drug: Mupirocin and Chlorhexidine

INTERVENTIONS:
Drug: Polyhexanide — Participants will apply Prontoderm® Nasal Gel and perform whole-body wash with Prontoderm® Foam daily for 5 days before surgery.
  Other Names: Prontoderm® Nasal Gel, Prontoderm® Foam
  Arms: Polyhexanide
Drug: Mupirocin and Chlorhexidine — Participants will apply Bactroban® Nasal ointment and perform whole-body wash with Lifo-Scrub® daily for 5 days before surgery.
  Other Names: Bactroban® Nasal Ointment, Lifo-Scrub®
  Arms: Mupirocin and Chlorhexidine

SUMMARY:
This pilot randomized controlled trial evaluates the feasibility, tolerability, and preliminary efficacy of a decolonization regimen using polyhexanide in reducing Staphylococcus aureus colonization in the preoperative phase of elective spine surgery, compared to the standard mupirocin and chlorhexidine regimen. The trial involves 24 participants randomized into two groups: one receiving polyhexanide and the other receiving mupirocin and chlorhexidine. The primary outcome is the randomization rate, with secondary outcomes including other feasibility outcomes, tolerability, and efficacy measures such as the reduction in S. aureus colony-forming units (CFUs) and changes in the nasal and skin microbiome composition.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Scheduled for elective spinal surgery
* Colonized with Staphylococcus aureus
* Informed consent provided

Exclusion Criteria:

* Emergency spine surgery
* Methicillin-resistant Staphylococcus aureus (MRSA) or mupirocin-resistant S. aureus
* Known allergies to products used in the trial
* Pregnant or breastfeeding women
* Recent antibiotic therapy (within 14 days)
* Known non-compliance, substance abuse, or psychological disorders
* Participation in another antimicrobial trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
randomization rate | at study completion, an average of 2 years.
  proportion of enrolled patients who were randomized

SECONDARY OUTCOMES:
positive screening rate | at study completion, an average of 2 years
  proportion of screened patients who were eligible
recruitment rate | at study completion, an average of 2 years
  proportion of eligible patients who were enrolled
retention rate | at study completion, an average of 2 years
  treatment-specific proportion of participants remaining in the trial
adherence rate | at study completion, an average of 2 years
  treatment-specific proportion of participants completing the treatment
trial burden | from start of treatment until last visit, up to 10 days
  NRS ranging from 0 - no burden to 10 very burdensome
tolerability of decolonization regimen | day 5 of treatment
  NRS ranging from 0 - well tolerable to 10 not tolerable
burden caused by side effects | day 5 of treatment
  numeric rating scale (NRS) ranging from 0 - no burden to 10 very burdensome
willingness to participate in future main trial | from start of treatment until last visit, up to 10 days
  NRS ranging from 0 - very unlikely to 10 very likely
Staphylococcus aureus colonization | pre-treatment (-30days to -10days before surgery), post-treatment (first day after treatment), the day of discharge (within 3 to 5 days after treatment)
  Staphylococcus aureus colony-forming units grown in cultures from nasal and skin swabs
The rate of mupirocin or oxacillin resistance | pre-treatment (-30days to -10 days before surgery)
  Proportion of Isolated Staphylococcus aureus Strains with Mupirocin or Oxacillin Resistance
The rate of treatment side effects | day 1-5 of treatment]
  signs and symptoms during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No